CLINICAL TRIAL: NCT01261923
Title: Pharmacokinetics of 9-cis-retinoic Acid (Alitretinoin, Toctino®) in Patients
Brief Title: Pharmacokinetics of 9-cis-retinoic Acid (Alitretinoin, Toctino®) in Patients With Hepatic Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Frederik Grønhøj, MD, University Hospital, Gentofte, Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: Eudra CT 2010-020212-11
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Hepatic Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency | interventions — Alitretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alitretinoin - Hepatic Insufficiency (Experimental): metabolism of 30 mg alitretinoin single dose in 8 patients with Hepatic Insufficiency
  Interventions: Drug: Alitretinoin
- Alitretinoin - Hepatic Insufficiency Controls (Experimental): metabolism of 30 mg alitretinoin single dose in 8 healthy controls.
  Interventions: Drug: Alitretinoin

INTERVENTIONS:
Drug: Alitretinoin — 30 mg capsule of 9-cis-retinoic-acid (9-cis-RA)(Alitretinoin, Toctino®)
  Other Names: 9-cis-retinoic-acid (9-cis-RA)(Alitretinoin, Toctino®)

SUMMARY:
This study aims to investigate whether liver patients may tolerate alitretinoin by comparing metabolism in 8 such patients with the metabolism in 8 healthy controls

DETAILED DESCRIPTION:
This study aims to investigate whether liver patients may tolerate alitretinoin.

Toctino (alitretinoin) is a vitamin A like substance that has proven effective in the treatment of specially hand eczema. The medicine is taken as capsules daily for up to 3 months. Toctino is currently only approved for patients with normal liver function, because it has never been studied how drug metabolism and excretion occurs in liver disease patients. This, however, the investigators want to examine in order to achieve an additional treatment for patients with severe hand eczema and concomitant liver disease.

The study is a collaboration between dermatology and medical department, Gentofte Hospital and University of Copenhagen, where blood and urine tests will be conducted. From the medical department, 8 patients diagnosed with liver disease will be recruited. Patients should only receive a single dose of Toctino (30 mg capsules). 20 blood samples and one urine sample will be taken over the next 24 hours (approximately 250-300 ml) to measure the concentration of Toctino in blood and urine. Moreover, the urine will be collected over 24 hours. Then the investigators will recruit an 8-person control group that is matched according to gender, age and weight. In this control group will take exactly the same samples. Based on determining concentrations in blood and urine will be able to mathematically calculate how Toctino is absorbed, distributed and excreted in liver disease patients in conjunction with a healthy control group. The study will therefore help to determine what dose of Toctino that would be preferable in liver disease patients.

The survey is estimated to be associated with a very low risk both for participating patients and control group. Toctino is an approved drug and side effects occur almost exclusively in long term treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Be medically stable for at least 1 month before the intake of 9-cis-RA.
2. There must be an ultrasound scan of liver and abdomen within the last 3 months (liver size, ascites).
3. In women of childbearing age, there must be a negative pregnancy test, while that to be used adequate contraception (the pill, coil or surgical sterilization) at least 1 month after taking the study medication.

Exclusion Criteria:

1. Clinically significant deviations in routine blood tests (hematology, electrolytes and kid-ney, urinalysis). Differences attributable to underlying liver disease are excluded.
2. Encephalopathy (> grade II)
3. Concomitant treatment with drugs predominantly metabolised in the liver by CYP3A4.
4. Clinically significant ECG changes, cardiovascular disease and AMI within the last 12 months
5. Affected renal function judged by Cockcroft-Gault formula.
6. Epilepsy or significant neurological disease that requires drug therapy.
7. History of cerebrovascular relapse
8. Esophagus bleeding
9. Severe ascites
10. HIV
11. Mental illness.
12. Active cancer
13. Pregnancy or pregnancy plan within 3 months.
14. Breastfeeding women.
15. Participation in other clinical projects.
16. Intake of clinical trial medication in the past month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-12; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The investigators wish to investigate whether the metabolism of alitretinoin differs between healthy controls and patients with moderate to severe hepatic disease | 2 years
  The metabolism of alitretinoin will be examined by measuring blood concentrations after time: 0 , ¼, ½, ¾, 1, 1¼, 1½, 2, 2½, 3, 3½, 4, 5, 6, 8, 10, 12 and 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Grønhøj, MD DMSci, Principal Investigator — Gentofte Hospital
Locations (1):
- Gentofte Hospital, Hellerup, Denmark